CLINICAL TRIAL: NCT06335875
Title: Brain Small Chain Fatty Acid Metabolism in Bipolar Disorder: Ketones
Acronym: BIPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00227568
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: ketone ester; ketogenic diet; brain imaging
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bipolar Disorder (Experimental): Participants will follow an intervention consisting of dietary changes and ketone ester supplementation for 90 +/- 10 days. The dietary changes are intended to reduce glycemic spiking and include: not consuming sweets, not consuming soda, replacing 'white' grains with whole grain alternatives, and reserving any fruit consumption for the end of meals. During the same time period, participants will consume the ketone ester supplement, consisting of 19 g Juvenescence Cognitive Switch™ (=12.5 g active C8-KE) diluted in water twice per day.
  Interventions: Dietary Supplement: Ketone Ester Beverage; Behavioral: Low Glycemic Index Diet

INTERVENTIONS:
Dietary Supplement: Ketone Ester Beverage — Participants will consume ketone ester (KE) beverage, consisting of 19 g (=12.5 g active C8-KE) of Juvenescence Cognitive Switch™ diluted in water, twice per day
  Other Names: Juvenescence Cognitive Switch™
Behavioral: Low Glycemic Index Diet — Participants will practice four dietary changes: 1. Not consuming sweets/candy, 2. Not consuming soda, 3. Replacing 'white' grains with complex carbohydrates such as brown rice or quinoa, and 4. Reserving any fruit consumption for the end of meals.
  Other Names: Ketogenic-mimicking Diet

SUMMARY:
Small exploratory open-label pilot study to assess supplementation of a ketone ester (Juvenescence) combined with a 'ketogenic-mimicking diet' as a potential therapy for persons with bipolar disorder.

DETAILED DESCRIPTION:
The overarching goal of this open-label, exploratory pilot study is to explore biomechanistic effects of exogenous ketone supplementation combined with a low glycemic diet (in effect, a 'ketogenic-mimicking diet') for patients with bipolar disorder. This represents a less restrictive metabolic intervention compared to a strict ketogenic diet while replicating two foundational elements of the ketogenic diet: low levels of glycemic/insulin signaling and high levels of circulating ketones. In addition to assessments of mood stability and global functioning, functional neuroimaging data will be obtained to better characterize the biomechanistic effects of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Able to provide informed consent
* Diagnosis of bipolar disorder, type I or II as determined primarily via medical/psychiatric documentation provided from mental health provider with patient consent
* Regular access to smart phone capable of syncing biometric wearable data collection
* If taking psychiatric medications, on stable regimen as defined by no medication changes for mood stabilizers and/or antipsychotics in prior 4 weeks

Exclusion Criteria:

* Inability to adhere to dietary changes as specified in protocol (e.g., not in control of food selection)
* History of moderate-to-severe traumatic brain injury, e.g. loss of consciousness > 10 min, neurologic sequela
* Evidence of large vessel stroke or mass lesion on previous MRI or MRI obtained during study
* History of significant GI disease (e.g., malabsorptive disorder, gastric cancer, intestinal resection)
* Pregnancy (as determined via urine pregnancy test at study initiation), if capable of becoming pregnant, or breastfeeding
* Unwilling to utilize birth control method during course of study (e.g., barrier contraception, oral contraceptive, IUD), if capable of becoming pregnant
* Currently receiving treatment with insulin (e.g., chronic pancreatitis, diabetes mellitus)
* History of mitochondrial disorder and/or significant uncontrolled metabolic/medical disorder
* Active/current illicit substance use (and/or consumption of >1 alcoholic beverages per day) - defined as using psychoactive medications not as prescribed or using illicit substances (as determined via urine drug screen and screening interview)
* Use of marijuana or THC products more than once monthly on average
* Subjects with contra-indications to MR imaging, including pacemakers or severe claustrophobia, and/or size incompatible with scanner gantry, e. g., men over 6 feet tall that weigh more than 250 lbs, men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs. Subjects of these weights or greater typically have difficult fitting into the fMRI scanner properly.
* Suicidal thoughts with plans or intentions, as assessed by C-SSRS
* Any other condition or criteria that would preclude safe and meaningful participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Change in blood beta-hydroxybutyrate level | After 90 +/- 10 days of intervention
  Keto-Mojo devices will be used to measure blood beta-hydroxybutyrate levels at baseline and after taking the supplement to assess both immediate and sustained effects on blood beta-hydroxybutyrate. Measurements taken at baseline, mid-intervention, and post-intervention will be compared and regressed to analyze associated changes.

SECONDARY OUTCOMES:
Change in blood glucose lability | After 90 +/- 10 days of intervention
  Continuous glucose monitoring (CGM) devices will be used to capture blood glucose lability, defined as frequency of glycemic spiking averaged per day. Baseline blood glucose lability and post-intervention blood glucose lability will be compared to analyze associated changes.
Change in neural network stability | After 90 +/- 10 days of intervention
  Functional Magnetic Resonance Imaging (fMRI) will be used to measure neural network stability (defined by correlations and anticorrelations among brain regions over time. Computed neural network stability after the supplementation/dietary change period will be compared to computed neural network stability at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Domino's Farms, Ann Arbor, Michigan
  - University Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT06335875/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT06335875/ICF_001.pdf